CLINICAL TRIAL: NCT03492073
Title: Effectiveness of an Individual Mindfulness-based Intervention for Cancer Patients in a Advanced Stage of the Disease and Their Relatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2017-12-04; First posted 2018-04-10 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2017-12

CONDITIONS: Cancer
Keywords: Mindfulness; Oncology; Cancer; Emotional distress; Quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Supportive Mindfulness-based Program (Experimental): The program is based on 15/20 minutes sessions of meditative practices in which can participate only the patients, only his/her caregiver, or both.
  Number of sessions is an independent outcome, because it depends on the number of days of hospitalization.
  Interventions: Behavioral: Emotional Supportive Mindfulness-based Program
- Emotional Supportive Program (Active Comparator): The program is based on 15/20 minutes sessions based on narrative therapy, in which the patient or his/her caregiver or both can talk about their emotions.
  Number of sessions is an independent outcome, because it depends on the number of days of hospitalization.
  Interventions: Behavioral: Emotional Supportive Program

INTERVENTIONS:
Behavioral: Emotional Supportive Mindfulness-based Program — Mindfulness training
  Arms: Emotional Supportive Mindfulness-based Program
Behavioral: Emotional Supportive Program — Narrative-orientated therapy.
  Arms: Emotional Supportive Program

SUMMARY:
The importance of emotional regulation interventions in cancer patients and primary caregivers is clearly established, since it helps them manage their emotions.

The aim of the study was to analyze the differential effect between two Emotional Support programs, one of them based on Mindfulness, and the other one Emotional Support as usual, on advanced cancer patients (stage III & IV) admitted to a Madrid Community Hospital La Paz and their relatives.

DETAILED DESCRIPTION:
It is clearly demonstrated that Emotional Regulation interventions are very important in cancer patients in any stage of the disease.

Great emotional burden has also been described in case of main caregivers and other relatives of the patients.

Diagnosis, treatment and survival of cancer patients are related to a complex set of stressors that have their own effects on the results of the treatments: activity daily life changes, social impairment, role changes, thought about the possibility of a relapse and possibility of death…

It has been elucidated that psychological interventions, as cognitive therapy or other types of psychotherapy, may improve the psychosocial outcomes (for example, quality of life).

During the last years, many researches have assessed the effect of Mindfulness interventions on cancer patients. Mindfulness is defined as the intention of paying full attention, moment to moment, to your experiences, without judgement.

Regular Mindfulness practice cultivates an acceptance state, improves emotional regulation strategies, improves quality of life, reduces rumination thinking, anxiety and depression.

The general aim of the present investigation is studying the effect of an Emotional Supportive based-mindfulness Program versus an Emotional Supportive Program (without Mindfulness component). Both programs are offered to cancer patients in an advanced stage of disease, admitted in the oncology section of the Hospital Universitario La Paz, and their relatives.

The investigator's hypothesis are:

* Both programs will reduce emotional distress, decreasing from 4 to 5 points out of 10 on average on the Distress thermometer (DT).
* Both interventions will improve moderately the score on Quality of Life measures (EORTC QLQ-15-PAL), obtaining 10-20 more points than at the initial assessment.
* Both interventions will reduce the emotional burden of the main caregiver (ZARIT short-form), obtaining a score under 17 points, which indicates "no familiar giving-up".
* Emotional Supportive based-Mindfulness Program will improve the scores on Philadelphia Mindfulness Scale (PHLMS) and acceptance, more than the Emotional Supportive Program will do.

The investigators will conduct a Randomized Controlled Trial with two treatment arms in an advanced-cancer patients sample of patients under hospitalization at Hospital Universitario La Paz, Madrid.

After all recollection of data is done, the investigators will conduct statistic analysis in order to accept or refuse our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Being in treatment in one of the Oncology units at Hospital Universitario La Paz.
* Capable of a minimum level of performance that allows intervention.
* The doctor responsible of the patient considers that the program will help the cancer patient and that the patient is capable to participate on it.
* Capable of understanding and giving his or her written informed consent.

Exclusion Criteria:

* Intellectual disability or cognitive impairment or dementia.
* Insufficient knowledge of the language to understand and participate on the intervention program.
* Serious mental illness in acute state at the moment of the beginning of the intervention.
* Autolytic ideas at the moment of the assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Mindfulness | At day one of the intervention
  Philadelphia Mindfulness Scale (PHLMS). Attention to the present moment and Acceptance.
Mindfulness | At the end of the six sessions(each session is every three days)
  Philadelphia Mindfulness Scale (PHLMS). Attention to the present moment and Acceptance.

SECONDARY OUTCOMES:
Quality of life. | At day one of the intervention
  Quality of life in advanced-cancer patients. (EORTC QLQ - C15-PAL).
Caregiver emotional burden. | At day one of the intervention
  Zarit. Emotional burden of the main caregiver. Impact of caring, interpersonal relationship and self-efficacy expectations.
Emotional distress | At day one of the intervention
  Distress thermometer (DT), scores from 1 to 10. Emotional distress.
Daily life Performance | At day one of the intervention
  Karnofsky Performance Status. It gives a measure of the dependency level of the patients, and the level of support that the cancer patient needs.
Number of sessions | At the end of the six sessions(each session is every three days)
  number of sessions of emotional support intervention or mindfulness emotional support intervention
Quality of life. | At the end of the six sessions(each session is every three days)
  Quality of life in advanced-cancer patients. (EORTC QLQ - C15-PAL).
Caregiver emotional burden. | At the end of the six sessions(each session is every three days)
  Zarit. Emotional burden of the main caregiver. Impact of caring, interpersonal relationship and self-efficacy expectations.
Emotional distress | At the end of the six sessions(each session is every three days)
  Distress thermometer (DT), scores from 1 to 10. Emotional distress.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodriguez Vega, Study Chair — Hospital Universitario La Paz. Universidad Autónoma de Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fallowfield L, Jenkins V. Psychosocial/survivorship issues in breast cancer: are we doing better? J Natl Cancer Inst. 2014 Nov 27;107(1):335. doi: 10.1093/jnci/dju335. Print 2015 Jan. PMID 25432407
- [Background] Hewitt M, Breen N, Devesa S. Cancer prevalence and survivorship issues: analyses of the 1992 National Health Interview Survey. J Natl Cancer Inst. 1999 Sep 1;91(17):1480-6. doi: 10.1093/jnci/91.17.1480. PMID 10469749
- [Background] Alfano CM, Rowland JH. Recovery issues in cancer survivorship: a new challenge for supportive care. Cancer J. 2006 Sep-Oct;12(5):432-43. doi: 10.1097/00130404-200609000-00012. PMID 17034679
- [Background] Fors EA, Bertheussen GF, Thune I, Juvet LK, Elvsaas IK, Oldervoll L, Anker G, Falkmer U, Lundgren S, Leivseth G. Psychosocial interventions as part of breast cancer rehabilitation programs? Results from a systematic review. Psychooncology. 2011 Sep;20(9):909-18. doi: 10.1002/pon.1844. Epub 2010 Sep 6. PMID 20821803
- [Background] Lotfi-Jam K, Carey M, Jefford M, Schofield P, Charleson C, Aranda S. Nonpharmacologic strategies for managing common chemotherapy adverse effects: a systematic review. J Clin Oncol. 2008 Dec 1;26(34):5618-29. doi: 10.1200/JCO.2007.15.9053. Epub 2008 Nov 3. PMID 18981466
- [Background] Carlson LE. Mindfulness-based interventions for physical conditions: a narrative review evaluating levels of evidence. ISRN Psychiatry. 2012 Nov 14;2012:651583. doi: 10.5402/2012/651583. Print 2012. PMID 23762768
- [Background] Gil F, Grassi L, Travado L, Tomamichel M, Gonzalez JR; Southern European Psycho-Oncology Study Group. Use of distress and depression thermometers to measure psychosocial morbidity among southern European cancer patients. Support Care Cancer. 2005 Aug;13(8):600-6. doi: 10.1007/s00520-005-0780-0. Epub 2005 Mar 11. PMID 15761700
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Gort AM, March J, Gomez X, de Miguel M, Mazarico S, Balleste J. [Short Zarit scale in palliative care]. Med Clin (Barc). 2005 May 7;124(17):651-3. doi: 10.1157/13074742. Spanish. PMID 15882512
- [Background] Cardaciotto L, Herbert JD, Forman EM, Moitra E, Farrow V. The assessment of present-moment awareness and acceptance: the Philadelphia Mindfulness Scale. Assessment. 2008 Jun;15(2):204-23. doi: 10.1177/1073191107311467. Epub 2008 Jan 9. PMID 18187399